CLINICAL TRIAL: NCT00005382
Title: Sources of Variability in Peak Expiratory Flow
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4287; R01HL051975 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2001-11

CONDITIONS: Asthma; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To provide information necessary for the development of standards for peak expiratory flow (PEF) test performance in populations studies.

DETAILED DESCRIPTION:
BACKGROUND:

While PEF has routinely been applied in the diagnosis and management of asthma, scientists were finding new applications for PEF as both a clinical and epidemiologic tool for following individuals with pulmonary diseases, studying the natural history of chronic obstructive pulmonary disease, and evaluating the impact of environmental exposures on lung function. Yet the standardization of the PEF measurement lagged behind its application.

The little attention paid to the performance characteristics of the PEF maneuver contrasted sharply with the efforts to standardize measurement procedures for FEV1 and FVC. The American Thoracic Society devoted a great deal of attention to studying these measures and published guidelines for the standardization of their measurement. These guidelines included detailed protocols for calibrating equipment, administering the tests, determining reproducibility, and interpreting results.

The research provided data on the optimal number of trials per test session, the difference between a PEF performed during a full forced expiratory effort and that resulting from a short blast, the impact of test supervision on test performance, and the reproducibility of the PEF measurement.

DESIGN NARRATIVE:

A baseline survey of ventilatory function was performed using spirometry. PEF was measured daily with a mini-Wright Peak Flow Meter over a period of several weeks in a study of 201 normals (staff, faculty and graduate students at the University of Massachusetts Lowell). Serial PEF data were collected on a group of mild asthmatics identified in a local occupational medicine clinic. Finally, performance characteristics were examined in serial PEF data from two existing occupational cohort studies.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-07; Study Completion 1998-05 (Actual)